CLINICAL TRIAL: NCT00003245
Title: Phase II Study of Irinotecan for the Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Irinotecan in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066124; MDA-DM-97182; NCI-T97-0103; DM97-182 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-09-24 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients with recurrent or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate and toxicity of irinotecan when administered to patients with recurrent or refractory non-Hodgkin's lymphoma.

OUTLINE: Patients are stratified by disease category (aggressive vs indolent vs mantle cell lymphoma). Patients with aggressive and indolent lymphoma are further stratified as to being refractory (no complete response (CR) or partial response (PR) to initial therapy) vs recurrent (CR or PR to initial therapy); i.e, the following subcategories are used:

* Stratum I:Refractory aggressive non-Hodgkin's lymphoma (NHL)
* Stratum II:Recurrent aggressive NHL
* Stratum III: Refractory indolent NHL
* Stratum IV: Recurrent indolent NHL
* Stratum V: Mantle cell NHL All patients receive irinotecan intravenously every 21 days. Patients achieving CR or PR receive 6 courses. Patients may receive bone marrow transplantation after at least 2 courses.

Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: This study will accrue 18 patients per stratum; if at least three patients respond, an additional 25 patients will be accrued for a total of 43 evaluable patients per stratum. The total number accrued will be 90-215 over a period of approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or refractory non-Hodgkin's lymphoma

  * First relapse requires histologic confirmation of relapse
* No CNS metastases
* No lymphomatous meningitis
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 15-75

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Unless due to lymphoma:

  * Platelet count at least 100,000/mm^3
  * Absolute granulocyte count at least 1,500/mm^3
  * Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver involvement)

Renal:

* Creatinine no greater than 2.0 mg/dL
* Baseline calcium less than 12 mg/dL

Cardiovascular:

* No myocardial infarction within 6 months
* No congestive heart failure requiring therapy

Other:

* No history of seizures
* No uncontrolled diabetes mellitus (i.e., random blood sugar of at least 250 mg)
* No other concurrent severe disease
* No uncontrolled infection
* HIV negative
* No psychoses
* No prior malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cancer of the cervix unless surgically treated and disease free for at least 5 years
* Not pregnant or lactating
* Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation

Chemotherapy:

* No more than 2 prior chemotherapy regimens for treatment of lymphoma
* No prior irinotecan, topotecan or aminocamptothecin
* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* Radiotherapy that is not a part of a combined-modality therapy is counted as a regimen (see Chemotherapy)

Surgery:

* Not specified

Other:

* No phenytoin, phenobarbital, or other antiepileptic prophylaxis

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1998-02-18 (Actual); Primary Completion 2004-07-30 (Actual); Study Completion 2004-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States